CLINICAL TRIAL: NCT00031629
Title: A Phase II Evaluation of Docetaxel and Gemcitabine Plus G-CSF in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Combination Chemotherapy and Filgrastim or Pegfilgrastim in Treating Patients With Recurrent or Persistent Cancer of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0131G; NCI-2012-02456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069206; GOG-0131G (Other: Gynecologic Oncology Group); GOG-0131G (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Docetaxel; Filgrastim; Granulocyte Colony-Stimulating Factor; Gemcitabine; pegfilgrastim

ARMS (1):
- Treatment (gemcitabine, docetaxel, G-CSF, pegfilgrastim) (Experimental): Patients receive gemcitabine IV over 90 minutes on days 1 and 8, docetaxel IV over 1 hour on day 8, and G-CSF SC on days 9-15 or pegfilgrastim SC on day 9 only. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Biological: Filgrastim; Drug: Gemcitabine Hydrochloride; Biological: Pegfilgrastim

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; Filgrastim-sndz; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim; Zarxio
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Biological: Pegfilgrastim — Given IV
  Other Names: Filgrastim SD-01; filgrastim-SD/01; HSP-130; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Colony-stimulating factors such as filgrastim or pegfilgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. This phase II trial is studying how well combination chemotherapy plus filgrastim or pegfilgrastim works in treating patients with recurrent or persistent cancer of the uterus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of docetaxel, gemcitabine, and filgrastim (G-CSF) or pegfilgrastim in patients with persistent or recurrent uterine leiomyosarcoma.

II. Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE:

Patients receive gemcitabine IV over 90 minutes on days 1 and 8, docetaxel IV over 1 hour on day 8, and filgrastim (G-CSF) subcutaneously (SC) on days 9-15 or pegfilgrastim SC on day 9 only. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 10-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uterine leiomyosarcoma

  * Recurrent or persistent disease that is refractory to curative therapy or established treatments
  * Must have received 1 prior chemotherapy regimen that may include high-dose therapy, consolidation, or extended therapy after surgical or nonsurgical assessment
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Lesions within a previously irradiated field allowed provided progression is documented or biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Ineligible for a high priority GOG protocol
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.1 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No active infection requiring antibiotics
* No motor or sensory neuropathy greater than grade 1
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No more than 1 prior non-cytotoxic (biologic or cytostatic) regimen (e.g., monoclonal antibodies, cytokines, or small-molecule signal transduction inhibitors) for recurrent or persistent disease
* At least 3 weeks since prior biologic or immunologic therapy for this disease
* See Disease Characteristics
* See Biologic therapy
* At least 3 weeks since prior chemotherapy and recovered
* No prior docetaxel or gemcitabine
* No other prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial regimens
* No prior chemotherapy for another malignancy that would preclude study
* At least 1 week since prior hormonal therapy for this disease
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* See Disease Characteristics
* Recovered from prior recent surgery
* At least 3 weeks since other prior therapy for this disease
* No concurrent amifostine or other protective agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of objective response | Up to 5 years
Frequency of severity of observed adverse effects assessed using CTC version 2.0 | Up to 5 years
  The frequency and severity of all toxicities are tabulated from submitted case report forms and summarized for review.

CONTACTS AND LOCATIONS:
Overall Officials: Martee Hensley, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States